CLINICAL TRIAL: NCT01774266
Title: Screening and Triage Test for Early Detection of Gastric Cancer
Brief Title: Detection of Methylated Reprimo in Plasma for Asymptomatic Gastric Cancer
Acronym: DEMRAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Ministerio de Salud de Chile (Unknown); Hoffmann-La Roche (Industry); Red Salud UC (Unknown)
Responsible Party: Sponsor
Other Study IDs: D09I1137; 11-156 (Other: CEI-MEDUC)
Record Dates: First submitted 2013-01-19; First posted 2013-01-23 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Early Gastric Cancer
Keywords: Gastric Cancer; DNA methylation; Reprimo; cell-free DNA; non-invasive
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and biopsy samples are collected
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Molina - Chile: Molina is one of the counties with the highest mortality rate of gastric cancer in Chile. Molina has a population of 40.000 hab mostly rural. Half of the population lives in Molina city and the other half in the suburbs. Molina is located near the Mountain Andes.

SUMMARY:
In this proposal the investigators aim to develop a commercial kit to be used in primary screening and non-invasive triage for early detection of gastric cancer. This kit will be cost-effective and more accessible to the general population. In addition, the investigators would like to expand our current patent already submitted to INAPI (National Institute for Intellectual Property) and propose royalties to biomedical diagnostic companies for the use of our product at international level.

DETAILED DESCRIPTION:
Gastric cancer is the first cause of death in Chile and the second worldwide. Currently, no screening methods are available for early detection of gastric cancer at population level. The only available test is serum levels of pepsinogen I/II for gastric atrophy, a precursor lesion only for intestinal type with low risk to progress to gastric cancer. The investigators' previous work, supported by FONDECYT (National Council for Research and Technology) and FONIS (National Council for Research and Development of Human Health) both from the Government of Chile led us to discover a potential biomarker for early detection of gastric cancer, Reprimo, a tumor suppressor gene related to p53 in the arrest of G2-M of the cell cycle (Clin Cancer Res. 2008;14:6264-9). Here, the investigators propose to evaluate plasmatic detection of Reprimo in conjunction with gastric atrophy markers and H.pylori detection to establish a novel screening and triage strategy for early detection of gastric cancer. The aims are i) to determine sensitivity and specificity for Reprimo in the detection of gastric cancer in a high-risk population evaluated by upper gastrointestinal endoscopy (1,000 males, 30-74 y.o. low income, symptomatic or asymptomatic) and ii) to characterize at clinical, pathological and molecular level cases of gastric cancer identified and non-identified by direct detection of Reprimo along with atrophy, H.pylori and clinical markers. With this information, the investigators will develop an algorithm for screening and triage evaluating predictive values of plasmatic detection of Reprimo versus atrophy & H.pylori detection and clinical data in a general population (3,000 male/female, 40-70 y.o.) from a high-risk area for gastric cancer in Chile. In this step the investigators will evaluate also acceptability, efficacy and efficiency of the proposed algorithm. In this proposal the investigators aim to develop a commercial kit to be used in primary screening and non-invasive triage for early detection of gastric cancer. This kit will be cost-effective and more accessible to the general population. In addition, the investigators would like to expand the investigators' current patent already submitted to INAPI and propose royalties to biomedical diagnostic companies for the use of the investigators' product at international level.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age 40-70 y.o.

Exclusion Criteria:

* Gastric Cancer
* Dyspepsia
* Bleeding disorders

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3000 population base study from rural area in south of Chile. This is area has one of the highest incidence of gastric cancer in the world (35/100.000).
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Early detection of gastric cancer | 2 years
  Increase the frequency of early detection rate of gastric cancer

SECONDARY OUTCOMES:
Monitoring progression of disease | 2 years
  In the case in which diagnoses of gastric cancer will be made, the result of treatment will be measure

OTHER OUTCOMES:
Detection of H.pylori and gastric atrophy | 2 years
  The rate of H.pylori detection and gastric atrophy based on serum levels of H.pylori and Pepsinogens I/II ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Santa Rosa de Molina, Molina, Maule Region, Chile

REFERENCES:
- [Background] Bernal C, Aguayo F, Villarroel C, Vargas M, Diaz I, Ossandon FJ, Santibanez E, Palma M, Aravena E, Barrientos C, Corvalan AH. Reprimo as a potential biomarker for early detection in gastric cancer. Clin Cancer Res. 2008 Oct 1;14(19):6264-9. doi: 10.1158/1078-0432.CCR-07-4522. PMID 18829507
- [Derived] Carrasco G, Corvalan AH. Helicobacter pylori-Induced Chronic Gastritis and Assessing Risks for Gastric Cancer. Gastroenterol Res Pract. 2013;2013:393015. doi: 10.1155/2013/393015. Epub 2013 Jul 29. PMID 23983680
- See also: search for project D09I1137 — http://www.conicyt.cl/fondef/